CLINICAL TRIAL: NCT03784521
Title: Efficacy of Intravenous In-line Filter in Patient Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 116064
Record Dates: First submitted 2018-11-30; First posted 2018-12-24 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: SIRS
Keywords: SIRS; In-line filtration; Cardiac surgery

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-line filtration (Experimental): For patients randomized to in-line filtration, in-line filters (Pall, Dreieich, Germany) are used for all intravenous access during operation and postoperative period in intensive care unit (ICU).
  Interventions: Device: In-line filtration
- Control (Active Comparator): For patients randomized to control group, All intravenous access is managed routinely according to local standard care without filtration during operation and postoperative period in ICU.
  Interventions: Device: Standard care

INTERVENTIONS:
Device: In-line filtration — In-line filtration is used during anesthesia and intensive care unit in study group to purify fluids administrations.
  Arms: In-line filtration
Device: Standard care — Patients are treated with standard intravenous solutions and vascular access management
  Arms: Control

SUMMARY:
The aim of this study is to demonstrated efficacy of in-line filtration to reduce systemic inflammatory response syndrome (SIRS) ,specific organ dysfunction and complications in adult cardiac surgery. 486 patients undergoing cardiac surgery for acquired heart disease are 1:1 randomized into in-line filtration (study group) and non-filtration (control group). The incidence of SIRS, complications, daily SOFA (sequential organ failure assessment) score are compared between groups.

DETAILED DESCRIPTION:
This clinical trial is performed at Ramathibodi hospital, Mahidol university in Bangkok, Thailand. The protocol has been approved by institutional ethical committee (ref. ID 11-60-64) with informed consent required for all patients.

The incidences of SIRS between the control and the filter group in pediatrics population from previous study were 35% and 25.2% respectively (risk difference -11.3%, 95% CI -21.8 to -0.5%). The author estimated the sample size of 486 randomized patients to give 80% power at the 10% significant level (alpha 0.1, beta 0.8).

Patients aged 18 years or older undergoing elective cardiac surgery for acquired heart disease (including isolated coronary artery bypass grafting (CABG), isolated valve surgery, combined valve surgery, or concomitant CABG and valve surgery) are randomized 1:1 into in-line filtration (study group) and non-filtration (control group).

For patients randomized to in-line filtration, in-line filters (Pall, Dreieich, Germany) are used for all intravenous access during operation and postoperative period in intensive care unit (ICU).

For patients randomized to control group, All intravenous access is managed routinely according to local standard care without filtration during operation and postoperative period in ICU.

Primary endpoint of this study is the incidence of SIRS after cardiac surgery. SIRS is diagnosed when patients have two or more of these criteria: 1.Heart rate >90/min, 2.Temperature >38 °C or <36 °C, 3.Respiratory rate >20/min or Paco2 <32 mm Hg (4.3 kPa), and 4.White blood cell count >12000/mm3 or <4000/mm3 or >10% immature band.

Secondary endpoints are complications as defined by Society of Thoracic Surgeons (STS) Adult Cardiac Surgical Database, daily SOFA score and organ dysfunction as defined by The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3).

Continuous data were reported as mean (standard deviation, SD) or median (interquartile range, IQR) and compared by independent sample t-test or the Mann-Whitney U test. Categorical variables were presented as frequency (%) and analyzed by chi-squared or Fisher's exact test. Statistical significance was defined as a P-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older undergoing elective adult cardiac surgery

Exclusion Criteria:

* Emergency surgery
* Patient who does not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of SIRS after cardiac surgery | SIRS is evaluated every 24 hours from immediate post-op to 96 hours postoperatively
  SIRS is diagnosed when patients have two or more of these criteria: 1.Heart rate >90/min, 2.Temperature >38 °C or <36 °C, 3.Respiratory rate >20/min or Paco2 <32 mm Hg (4.3 kPa), and 4.White blood cell count >12000/mm3 or <4000/mm3 or >10% immature band.

SECONDARY OUTCOMES:
Daily SOFA score | SOFA score is evaluated every 24 hours from immediate post-op to 96 hours postoperatively
  Daily SOFA score and organ dysfunction are as defined by The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each organ has a possible dysfunction score of 0 to 4.
Incidence of Operative mortality | up to 1 month postoperatively
  Operative mortality includes both (1) all deaths occurring during the hospitalization in which the operation was performed, even if after 30 days; and (2) those deaths occurring after discharge from the hospital, but within 30 days of the procedure.
Incidence of Permanent Stroke | up to 1 month postoperatively
  Postoperative stroke (i.e., any confirmed neurological deficit of abrupt onset caused by a disturbance in blood supply to the brain that did not resolve within 24 hours.
Incidence of Renal Failure | up to 1 month postoperatively
  Acute or worsening renal failure resulting in one or more of the following:
  1. Increase of serum creatinine to ≥ 4.0 with an increase of at least 0.5mg/dl or 3x most recent preoperative creatinine level.
  2. A new requirement for dialysis postoperatively.
Incidence of Prolonged Ventilation > 24 hours | up to 1 month postoperatively
  Prolonged post-operative pulmonary ventilation > 24.0 hours. The hours of postoperative ventilation time include OR exit until extubation, plus any additional hours following reintubation.
Incidence of Deep sternal wound infection | up to 1 month postoperatively
  Deep sternal wound infection or mediastinitis (according to CDC definition) diagnosed within 30 days of the operation or any time during the hospitalization for the surgery.
Incidence of Reoperation for any reason | up to 1 month postoperatively
  Reoperation for bleeding/tamponade, valvular dysfunction, graft occlusion, other cardiac reason, or non-cardiac reason
Incidence of Major Morbidity or Operative Mortality | up to 1 month postoperatively
  A composite endpoint defined as any of the outcomes listed above, including; Operative mortality, Permanent Stroke, Renal Failure, Prolonged Ventilation > 24 hours, Deep sternal wound infection, Reoperation for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Narongrit Kantathut, MD, Principal Investigator — Ramathibodi hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sasse M, Dziuba F, Jack T, Koditz H, Kaussen T, Bertram H, Beerbaum P, Boehne M. In-line Filtration Decreases Systemic Inflammatory Response Syndrome, Renal and Hematologic Dysfunction in Pediatric Cardiac Intensive Care Patients. Pediatr Cardiol. 2015 Aug;36(6):1270-8. doi: 10.1007/s00246-015-1157-x. Epub 2015 Apr 7. PMID 25845941